CLINICAL TRIAL: NCT02743741
Title: A Prospective Single-Arm, Multi-Centre, Study of the Efficacy and Safety of Lutetium-177 Octreotate (Lu-DOTATATE) Treatment With Individualized Dosimetry in Patients With 68Ga-DOTATATE Identified Somatostatin Receptor Positive Neuroendocrine Tumors
Brief Title: Lu-DOTATATE Treatment in Patients With 68Ga-DOTATATE Somatostatin Receptor Positive Neuroendocrine Tumors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Ozmosis Research Inc. (Industry); Cancer Care Ontario (Other); Canadian Molecular Imaging Probe Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-067
Record Dates: First submitted 2016-04-13; First posted 2016-04-19 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Neuroendocrine Tumors
Keywords: Somatostatin Receptor Positive Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lutetium-177 Octreotate (Experimental): Lutetium-177 Octreotate 200 mCi (7.4 GBq) by IV for 18-30 weeks
  Interventions: Drug: Lutetium-177 Octreotate

INTERVENTIONS:
Drug: Lutetium-177 Octreotate — Radiopharmaceutical
  Other Names: Lu-DOTATATE; [Lu-177]-DOTATATE

SUMMARY:
This is a prospective single arm, multicenter study will evaluate the efficacy and safety of Lutetium-177 Octreotate in patients with neuroendocrine tumors who has positive Somatostatin receptor identified by 68Ga-DOTATATE. 195 patients will be enrolled totally. Patient who has progressed with neuroendocrine tumor will be evaluated by the tumor board first and eligible patients will undergo diagnostic Ga 68 PET scan. Patients who showed Somatostatin will undergo 4 cycles of Lu-DOTATATE treatment. Dose adjustment for Cycle 2-4 will be made based on individualized dosimetry, as well as creatinine clearance and hematological parameters. Patients will be evaluated progression free survival at 12 months from last dose. Patients who are negative for somatostatin will not receive 68Ga-DOTATATE treatment but will be followed until progression and acts as control group.

ELIGIBILITY:
Please note that only Ontario residents will be eligible for participation in this trial.

Inclusion Criteria:

1. Biopsy-proven neuroendocrine tumor
2. ECOG performance status ≤ 2
3. Ki-67 index ≤ 30%
4. Evidence of progressive disease demonstrated by imaging within six months prior to study enrollment as defined by RECIST v1.1.

   * Tumor board discussion of cases to confirm suitability for participation in the clinical trial is required. Review should include but not limited to imaging review, pathology (including Ki 67) and treatment options.
   * Patients with objective evidence (imaging, or biochemical) that is insufficient to be classified by RECIST 1.1 criteria can be eligible if after provincial multidisciplinary tumor board discussion a consensus for progression eligibility is reached.
   * The tumor board would consider exemptions if the magnitude of change is adequate by other definitions (e.g. using structural and contrast patterns and biochemical changes).
   * Where clinically indicated, formal consultation on pathology, diagnostic imaging to facilitate criteria assessment (including 68Ga PET performed as part of the diagnostic procedure) is strongly recommended.
5. Adequate lab parameters within 2 weeks prior to enrollment:

   * Serum creatinine ≤ 150 μmol/L
   * Calculated CrCl or measured GFR ≥ 30 mL/min (measured GFR may be done within 4 weeks prior to enrollment)
   * Haemoglobin ≥ 90 g/L
   * WBC ≥ 2 x 109/L
   * Platelets ≥ 100 x 109/L
6. Adequate liver function tests within 2 weeks prior to enrollment:

   * total bilirubin ≤ 5 x ULN
   * ALT ≤ 5 x ULN
   * AST ≤ 5 x ULN
   * alkaline phosphatase ≤ 5 x ULN
7. Signed informed consent
8. Patients with extensive bone metastases (e.g. >25% of bone marrow involvement are eligible but requires careful monitoring of hematological reserve
9. Subject's willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
10. Age ≥ 18 years.

Exclusion Criteria:

1. Life expectancy <12 weeks
2. An option for curative surgical or medical therapy or local liver embolization is feasible
3. Candidate for curative and/or debulking surgical resections
4. Systemic, biologic, other radioisotope, embolization therapies within ≤4 weeks prior to the first dose of 177Lu.
5. Prior radiotherapy to target lesion(s) within ≤12 weeks prior to study enrollment [radiotherapy to non-target lesions permitted].
6. Prior therapy with any systemic radionuclide therapy.
7. Radiotherapy to more than 25% of the bone marrow.
8. Known brain metastases (unless metastases have been treated and are stable for ≥ 6 months).
9. Uncontrolled diabetes mellitus
10. Co-morbidities that may interfere with delivery of 177Lu (e.g. urinary incontinence).
11. Second cancer(s) with clinical or biochemical progression within the last 3 years.
12. Pregnancy or breast feeding. Female subjects must be surgically sterile or postmenopausal, or must agree to use effective contraception during the period of therapy. All female subjects with reproductive potential must have a negative pregnancy test (serum) prior to enrolment. Male subjects must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate
13. Other condition, illness, psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation, 68Ga or 177Lu administration, or may interfere with the interpretation of study results and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients progression-free using RECIST 1.1 criteria | Up to 12 months

SECONDARY OUTCOMES:
The overall response rate as determined by structural imaging using RECIST criteria. | Up to 5 years
The biochemical response rate (as defined by biochemical responses: serum chromogranin A and 24 hr urinary 5HIAA). | Up to 5 years
The acute and late adverse effects of Lu-DOTATATE (177Lu) using CTCAE Version 4.03 | Up to 5 years
Overall survival | Up to 5 years
The Quality of Life (QoL) in patients treated with Lu-DOTATATE (177Lu) | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sunnybrook Odette Cancer Center, Toronto, Ontario